CLINICAL TRIAL: NCT02926508
Title: Investigating the Effects of a Prebiotic Supplement on Learning and Behaviour in Children From Academic Year Groups 3, 4 and 5, Whose Reading Scores Suggest There is Room for Improvement: a Randomised Placebo-controlled Study
Brief Title: Oxford Study of Prebiotics in Children
Acronym: OxPiC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Oxford (Other)
Collaborators: Clasado Biosciences Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: R44843/RE001
Record Dates: First submitted 2016-08-18; First posted 2016-10-06 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Behaviour
Keywords: Reading; Learning; Cognition
MeSH Terms: conditions — Behavior | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prebiotic (Bimuno) (Experimental): Bimuno (B-GOS, Galacto-oligosaccharides, produced and provided by Clasado BioSciences Ltd)
  Interventions: Dietary Supplement: Bimuno (BGOS)
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Bimuno (BGOS) — The active supplement of the food supplement (Bimuno) used in this study is called galacto-oliogosaccharides (Bimuno®, BGOS). BGOS is a compound metabolised by specific bifidobacteria, which are beneficial bacteria, in our colon. Bimuno (2.3 calories) is composed by the following ingredients per gram of Bimuno: 0.96g dry matter; <01g Fat; <0.06g Protein; 0.821g GOS; 0.119g Lactose; 0.0331g Glucose and 0.0029g Galactose. Bimuno is tasteless.
  Bimuno will be supplied in coded sachets (3.5g) for dispensing by parents. Each participant will be required to consume 1 sachet daily during breakfast, by mixing it with food or in a drink.
  Arms: Prebiotic (Bimuno)
Other: Maltodextrin — Maltodextrin is a polysaccharide in powder form, which grows most bacteria in the gut, and not specifically the beneficial bifidobacteria.
  The placebo will also be provided in daily coded sachets (3.5g) for dispensing by parents. Each participant will be required to consume 1 sachet daily during breakfast, by mixing it with food or in a drink.
  This placebo has been used in previous studies, in which Bimuno was used as the active intervention. The placebo will be similar in taste and colour to the active intervention.
  Arms: Placebo

SUMMARY:
Recently, there has been an emerging interest in how manipulating gut microbiota (which is composed by microorganisms living in our digestive system) can influence learning, memory and cognition. This influence is thought to primarily occur via the gut endocrine and immune systems, and the vagus nerve, all of which influence brain function and are modulated by intestinal microorganisms. One way to manipulate the microbiota is to ingest dietary compounds, such as prebiotics.

Prebiotics are non-digestible dietary fibres that enhance the growth of "healthy" bacteria in the intestines when given in adequate amounts. Prebiotics are relatively stable, can be stored at room temperature and can be easily added to foods or drinks. They are not degraded by enzymes and acids in the digestive tract; therefore they reach the colon relatively unchanged, where they are metabolised by specific bacteria, thus promoting their beneficial effects. Prebiotics can be found in very small proportions in vegetables and fruits such as leeks, onions, tomatoes, garlic, etc., but this naturally occurring quantity is generally insufficient to promote a significant growth of beneficial bacteria. Therefore, large quantities of purified prebiotics are available as powder supplements and sold in packages of the appropriate dose.

Pre-clinical studies in animals have shown that prebiotics modulates brain expression of key molecules involved in cognition and brain health in rats. These findings therefore highlight the potential of influencing cognition through the manipulation of gut microbiota (in this case, via the ingestion of a prebiotic).

Building on this evidence, the aim of this study is to investigate how manipulating gut microbiota can influence reading, learning and behaviour in a group of children whose reading scores suggest there is room for improvement.

DETAILED DESCRIPTION:
This study has a randomised, double-blind, between-subjects, placebo-controlled design, whereby participants will receive a 12-week treatment with Bimuno or a matched placebo.

Children whose Key Stage 1 scores indicate they are within the lowest quintile for literacy, but whose teachers do not judge them to have any other significant learning difficulties, will be invited to be screened for the study. The teacher will also need to confirm if their reading is still a cause of concern; if not, the children will no longer be considered for inclusion in the study. Teachers will be asked to add the names of any additional children whose reading shows room for improvement. These children will be assessed to ensure they meet inclusion/exclusion criteria.

If the child passes this initial school screening stage, and conditional to parental consent, he/she will then be assessed using the reading test from the British Ability Scale (BAS). Only those whose reading falls into the bottom 34th centile on the BAS word reading measure will be invited to take part in the full study.

The study will include three sessions in total (all taking place at schools): (1) screening session, (2) baseline session and (3) post-intervention testing session. Children will also be asked to wear an actigraphy device for 5 consecutive nights before and after the treatment. In addition, children will be asked to give saliva samples on a few occasions (both at home - pre- and post-intervention -, as well as during the baseline and testing session visits).

Parents and teachers will be asked to complete standardised questionnaires also before and after the treatment ends.

ELIGIBILITY:
Inclusion Criteria:

Children

* Children from academic year groups 3, 4 and 5 (who are generally aged 7 to 9 years), male or female, who are underperforming in literacy skills according to nationally standardised assessments of scholastic achievement at age 7 (Key Stage 1). To be eligible, children must be confirmed to score ≤ 34th centile for reading, but are not judged by their teachers to have any other significant learning difficulties;
* Children are willing and able to give informed assent for participation in the study and to comply with all study requirements;
* Fluent English speakers only, as the measures have only been validated on such children.

Parents

* Parents of those children selected to do the study (after doing the screening reading test), and who are willing and able to give informed consent and to comply with all study requirements;
* Fluent English speakers only, as the measures have only been validated on such adults.

Teachers

• Primary school teachers of children who are selected to do the study, and who are willing and able to give informed consent and to comply with all study requirements.

Exclusion Criteria:

Children

* Major learning disabilities or medical disorders (including diseases affecting the human gastrointestinal tract);
* Participants who are currently taking (or intending to take) any medication that may affect the outcomes, including medications affecting brain processing, sedation, gut health and motility (examples include antidepressants, anxiolytics, cholinergic agonists, among others);
* Participants who have a known intolerance to lactose;
* Participants who are taking any other food supplements which, in the opinion of the Investigators, may affect the results;
* Antibiotic, probiotic and/or prebiotic treatment in at least the 2 previous months;
* Any significant change in diet which, to the discretion of the Investigators, may affect the results;
* Participants who have recently participated in another research trial which, to the discretion of the Investigators, may affect the results;
* Any firm plans of the child and family to move schools during the intervention period;
* Any other significant finding arising during the screening/selection process which, in the opinion of the Investigators, may influence the participant's ability to take part in the study or the study results.

Parents • Lack of availability to comply with study procedures.

Teachers

• Lack of availability to comply with study procedures.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
British Ability Scale (BAS) II Word Scale | 12 weeks
British Ability Scale (BAS) Digit Span Scale | 12 weeks
CogTrack Precision Cognitive Tests | 12 weeks

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory for children - child's version | 12 weeks
State-Trait Anxiety Inventory for children - parent's version | 12 weeks
Mood and Feelings Questionnaire - child's version | 12 weeks
Mood and Feelings Questionnaire - parent's version | 12 weeks
Child Sleep Habits Questionnaire (CSHQ) | 12 weeks
Objective sleep as measured by actigraphy | 12 weeks
Gastro-intestinal function diary | 12 weeks
Sleep diary | 12 weeks
Conners Teacher Rating Scale (CTRS-L) | 12 weeks
Conners Parent Rating Scale (CPRS-L) | 12 weeks
Saliva samples (to measure cortisol and immune markers) | 12 weeks
School attendance | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Department of Psychiatry, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided